CLINICAL TRIAL: NCT02543346
Title: Comparability and Standardization of Controlled Allergen Challenge Facilities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Biogenics Research Chamber, LLC (Industry)
Responsible Party: Principal Investigator, Dr. Anne Ellis, Chair, Division of Allergy & Immunology, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EEU-BRC-001
Record Dates: First submitted 2015-09-02; First posted 2015-09-07 (Estimated); Results first posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Cetirizine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- cetirizine hydrochloride (Other)
  Interventions: Drug: Cetirizine
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Cetirizine — Participants will receive either cetirizine (10mg tablet, orally) or a placebo (sugar pill) at one of the two treatment visits.
  Other Names: Zyrtec; Reactine
  Arms: cetirizine hydrochloride
Other: Placebo — Participants will receive either a placebo or cetirizine (10mg tablet, orally) at one of the two treatment visits
  Arms: placebo

SUMMARY:
Allergen challenge facilities have been utilized for many years in clinical drug trials studying onset of action, proof of concept, duration of action, and efficacy. Each facility has somewhat different design characteristics and pollen dispersal technologies. Facilities are located in disparate geographic areas and have populations of participants who are sensitized to allergens unique to that area. Therefore, facilities have operated as single sites with little effort to evaluate facility comparability or to attempt standardization across facilities. The purpose of this study is to compare the two sites and assess whether the sites are able to achieve similar symptom scores.

DETAILED DESCRIPTION:
When CACF have been designed with a high degree of rigor, quality assurance and validation testing, the exposure to controlled levels of pollen in such facilities as the Environmental Exposure Unit (EEU) and the Biogenics Research Chamber (BRC) will demonstrate comparable/standardized symptomatic responses. This will be demonstrable not only following pollen exposure but will also have similar reductions in symptoms following treatment with a Food and Drug Administration (FDA) approved medication known to be effective for the treatment of seasonal allergic rhinoconjunctivitis ( SAR); cetirizine 10mg. Because of quality assurance and validation testing completed at these facilities a priori, this comparability will be demonstrated despite their disparate geographical physical locations and the utilization of these facilities of somewhat different mechanical and technical materials and methods to achieve similar outcomes.

This multi-center study of SAR will enroll 50 participants at each site. These participants will be age 18-65, male and female, with a mixture of ethnic groups. The study will involve 3 Phases: Screening, Treatment Exposure Visit, and a cross-over Treatment Exposure Visit. In all stages, a CACF visit will be pivotal to determine participant eligibility for enrollment and response to therapy. The qualifying participants will receive a double-blinded, placebo-controlled, crossover intervention with cetirizine HCl 10mg.

All participants will give written informed consent prior to any study related procedures being performed. Participants who meet all inclusion/exclusion criteria during the screening process will be asked to return to the EEU for their first pollen exposure visit (Treatment Visit #1). At the Screening Visit participants will provide a full medical history and undergo a physical examination. They will have their height/weight and vitals measured and skin testing will be performed to confirm allergic response to a panel of common aeroallergens. Women of child bearing potential will undergo a urine pregnancy test to rule out pregnancy. Eligible participants will be invited back to the research centre for 4 pollen exposure visits at 2 of these visits participants will receive either cetirizine or placebo. All participants will receive placebo at some point throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* history of rhinoconjunctivitis during ragweed season for a minimum of 2 years, including the previous 2 ragweed seasons.
* positive skin test to ragweed allergen.

Exclusion Criteria:

* participant is pregnant, lactating or actively trying to conceive.
* has a history of receiving immunotherapy containing short ragweed within the last 3 years.
* participant has current allergy symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Ellis, MD, Principal Investigator — Queen's University
Locations (2):
- Biogenics Research Chamber, San Antonio, Texas, United States
- Kingston General Hospital, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 149 individuals were screened across both study sites; 78 individuals were screened at the Environmental Exposure Unit in Kingston, Ontario, Canada. 71 individuals were screened at the Biogenics Research Chamber in San Antonio, Texas, USA.
Pre-assignment Details: A total of 98 of 149 individuals were randomized (51 individuals for the Environmental Exposure Unit, 47 individuals for the Biogenics Research Chamber). Of those not randomized, 5 did not meet inclusion criteria, and 46 were discontinued prior to randomization due to not meeting eligibility criteria.
Groups:
- EEU: Cetirizine First, Then Placebo: At the EEU, participants attended the first priming visit. At least 3 days later, participants attended the first treatment visit (5-h pollen exposure) and received one Cetirizine 10 mg tablet at the 150-min time point. After a washout period of at least 14 days, participants attended the second priming visit. At least 3 days later, participants attended the second treatment visit (5-h pollen exposure) and received one matching placebo tablet at the 150-min time point.
- EEU: Placebo First, Then Cetirizine: At the EEU, participants attended the first priming visit. At least 3 days later, participants attended the first treatment visit (5-h pollen exposure) and received one matching placebo tablet at the 150-min time point. After a washout period of at least 14 days, participants attended the second priming visit. At least 3 days later, participants attended the second treatment visit (5-h pollen exposure) and received one Cetirizine 10 mg tablet at the 150-min time point.
- BRC: Cetirizine First, Then Placebo: At the BRC, participants attended the first priming visit. At least 3 days later, participants attended the first treatment visit (5-h pollen exposure) and received one Cetirizine 10 mg tablet at the 150-min time point. After a washout period of at least 14 days, participants attended the second priming visit. At least 3 days later, participants attended the second treatment visit (5-h pollen exposure) and received one matching placebo tablet at the 150-min time point.
- BRC: Placebo First, Then Cetirizine: At the BRC, participants attended the first priming visit. At least 3 days later, participants attended the first treatment visit (5-h pollen exposure) and received one matching placebo tablet at the 150-min time point. After a washout period of at least 14 days, participants attended the second priming visit. At least 3 days later, participants attended the second treatment visit (5-h pollen exposure) and received one Cetirizine 10 mg tablet at the 150-min time point.
Period: First Priming Visit
Arm/Group | EEU: Cetirizine First, Then Placebo | EEU: Placebo First, Then Cetirizine | BRC: Cetirizine First, Then Placebo | BRC: Placebo First, Then Cetirizine
Started | 26 | 25 | 24 | 23
Completed | 26 | 25 | 24 | 23
Not Completed | 0 | 0 | 0 | 0
Period: First Treatment Visit
Arm/Group | EEU: Cetirizine First, Then Placebo | EEU: Placebo First, Then Cetirizine | BRC: Cetirizine First, Then Placebo | BRC: Placebo First, Then Cetirizine
Started | 26 | 25 | 24 | 23
Completed | 26 | 25 | 24 | 23
Not Completed | 0 | 0 | 0 | 0
Period: Washout (at Least 14 Days)
Arm/Group | EEU: Cetirizine First, Then Placebo | EEU: Placebo First, Then Cetirizine | BRC: Cetirizine First, Then Placebo | BRC: Placebo First, Then Cetirizine
Started | 26 | 25 | 24 | 23
Completed | 26 | 25 | 24 | 23
Not Completed | 0 | 0 | 0 | 0
Period: Second Priming Visit
Arm/Group | EEU: Cetirizine First, Then Placebo | EEU: Placebo First, Then Cetirizine | BRC: Cetirizine First, Then Placebo | BRC: Placebo First, Then Cetirizine
Started | 26 | 25 | 24 | 23
Completed | 25 | 23 | 22 | 21
Not Completed | 1 | 2 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Second Treatment Visit
Arm/Group | EEU: Cetirizine First, Then Placebo | EEU: Placebo First, Then Cetirizine | BRC: Cetirizine First, Then Placebo | BRC: Placebo First, Then Cetirizine
Started | 25 | 23 | 22 | 21
Completed | 25 | 23 | 22 | 21
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes participants at both EEU and BRC sites who were randomized to receive both interventions (Cetirizine 10 mg and Placebo).
Groups:
- All Study Participants: Includes all participants at the EEU and BRC sites. All participants were randomized to receive both interventions (Cetirizine 10 mg and Placebo).
Arm/Group | All Study Participants
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 71

OUTCOME MEASURES:

1. Primary Outcome: Comparison of TRSS From Baseline Between the EEU and BRC in the Cetirizine 10 mg and Placebo Groups.
Description: Participants recorded their nasal and ocular symptoms at baseline and during the intervention visits.
  The TRSS is a composite score comprised of 4 nasal (runny nose, sneezing, nasal itch, nasal congestion) and 3 ocular (itchy eyes, watery eyes, red/burning eyes) symptoms. The severity of each individual symptom is rated on a 4-point scale (0 to 3) and are summed for a maximum TRSS of 21 (0 to 21).The 4-point scale includes a severity score of 0 (None: no sign/symptom is evident), 1 (Mild: Sign/symptom clearly present, but minimal awareness; easily tolerated), 2 (Moderate: Definite awareness of sign/symptom that is bothersome, but tolerable), 3 (Severe: Sign/symptom that is hard to tolerate; causes interference with activities during the challenge session. A higher score indicates higher symptom severity.
Time Frame: First treatment visit and second treatment visit.
Population: Efficacy analyses included all randomized participants who received at least 1 dose of study medication (Cetirizine 10 mg or Placebo).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | EEU Placebo | BRC Placebo | EEU Cetirizine | BRC Cetirizine
Number analyzed (Participants) | 48 | 43 | 48 | 43
score on a scale | 11.9 (0.49) | 11.7 (0.51) | 11.5 (0.49) | 10.8 (0.52)

2. Secondary Outcome: Comparison of TNSS From Baseline Between the EEU and BRC in the Cetirizine 10 mg and Placebo Groups.
Description: Participants recorded their nasal and ocular symptoms at baseline and during the intervention visits.
  The Total Nasal Symptom Score (TNSS) is a composite score comprised of 4 nasal (runny nose, sneezing, nasal itch, nasal congestion) symptoms. The severity of each individual symptom is rated on a 4-point scale (0 to 3) and are summed for a maximum TNSS of 12 (0 to 12) .The 4-point scale includes a severity score of 0 (None: no sign/symptom is evident), 1 (Mild: Sign/symptom clearly present, but minimal awareness; easily tolerated), 2 (Moderate: Definite awareness of sign/symptom that is bothersome, but tolerable), 3 (Severe: Sign/symptom that is hard to tolerate; causes interference with activities during the challenge session. A higher score indicates higher symptom severity.
Time Frame: First treatment visit and second treatment visit.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | EEU Placebo | BRC Placebo | EEU Cetirizine | BRC Cetirizine
Number analyzed (Participants) | 48 | 43 | 48 | 43
score on a scale | 7.3 (0.30) | 7.5 (0.32) | 7.1 (0.30) | 6.9 (0.32)

3. Secondary Outcome: Comparison of TOSS From Baseline Between the EEU and BRC in the Cetirizine 10 mg and Placebo Groups.
Description: Participants recorded their nasal and ocular symptoms at baseline and during the intervention visits.
  The Total Ocular Symptom Score (TOSS) is a composite score comprised of 3 ocular (itchy eyes, watery eyes, red/burning eyes) symptoms. The severity of each individual symptom is rated on a 4-point scale (0 to 3) and are summed for a maximum TOSS of 9 (0 to 9) .The 4-point scale includes a severity score of 0 (None: no sign/symptom is evident), 1 (Mild: Sign/symptom clearly present, but minimal awareness; easily tolerated), 2 (Moderate: Definite awareness of sign/symptom that is bothersome, but tolerable), 3 (Severe: Sign/symptom that is hard to tolerate; causes interference with activities during the challenge session. A higher score indicates higher symptom severity.
Time Frame: First treatment visit and second treatment visit.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | EEU Placebo | BRC Placebo | EEU Cetirizine | BRC Cetirizine
Number analyzed (Participants) | 47 | 43 | 47 | 43
score on a scale | 4.6 (0.23) | 4.2 (0.24) | 4.4 (0.23) | 3.9 (0.24)

4. Secondary Outcome: Comparison of GRCS From Baseline Between the EEU and BRC in the Cetirizine 10 mg and Placebo Groups.
Description: Participants recorded how they were feeling at baseline and at the end of both treatment visits.
  The Global Rating of Change Scale documents the changes in the participant's emotions. The scale ranges from +7 (A very great deal better) to -7 (A very great deal worse) with 0 being no change. A higher score indicates a better outcome.
Time Frame: First treatment visit and second treatment visit.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | EEU Placebo | BRC Placebo | EEU Cetirizine | BRC Cetirizine
Number analyzed (Participants) | 48 | 43 | 48 | 43
score on a scale | 1.2 (0.55) | -0.1 (0.57) | 1.8 (0.55) | 0.9 (0.58)

5. Secondary Outcome: Comparison of VAS From Baseline Between the EEU and BRC in the Cetirizine 10 mg and Placebo Groups.
Description: Participants recorded the severity of all nasal and ocular symptoms at baseline and at the end of both treatment visits.
  The Visual Analogue Scale (VAS) is a single overall rating of the severity of all nasal and ocular symptoms experienced by the participant. The scale ranges from 0 to 100 mm with 0 mm being no symptoms and 100 mm being the worst symptoms the participant has ever felt.
Time Frame: First treatment visit and second treatment visit.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | EEU Placebo | BRC Placebo | EEU Cetirizine | BRC Cetirizine
Number analyzed (Participants) | 48 | 43 | 48 | 43
units on a scale | 52.7 (3.98) | 47.7 (4.18) | 45.3 (4.00) | 44.1 (4.19)

ADVERSE EVENTS:
Time Frame: Collection of adverse event data started after the first dose of study medication (Cetirizine 10 mg or Placebo) until study completion, a duration of 1 month.
Description: The evaluable population included all participants who were randomized. This includes 51 participants in the EEU and 47 participants in the BRC.
Groups:
- EEU Placebo: Participants in the EEU who received one matching placebo at either the first or second treatment visit.
- BRC Placebo: Participants in the BRC who received one matching placebo at either the first or second treatment visit.
- EEU Cetirizine: Participants in the EEU who received Cetirizine at either the first or second treatment visit.
- BRC Cetirizine: Participants in the BRC who received Cetirizine at either the first or second treatment visit.
Arm/Group | EEU Placebo | BRC Placebo | EEU Cetirizine | BRC Cetirizine
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/47 | 0/51 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/47 | 0/51 | 0/47
Other Adverse Events (participants affected / at risk) | 0/51 | 0/47 | 0/51 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No